CLINICAL TRIAL: NCT00178152
Title: The Implication of Erythema Toxicum Neonatorum in Newborns on the Development of Future Asthma
Brief Title: Erythema Toxicum Neonatorum in Newborns and the Development of Asthma
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Jill S. Halterman, MD, MPH, University of Rochester
Other Study IDs: 11627
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Asthma; Erythema Toxicum Neonatorum
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Erythema Toxicum Neonatorum (ETN) is a common skin finding that affects healthy full-term babies. Several authors have commented on the possible relationship between ETN and the development of atopic conditions, such as atopic dermatitis or respiratory disease later in life. There is a paucity of research addressing this issue.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3-9 years who have had at least 2 asthma diagnoses within the last 2 years.
* Control subjects will be age matched and without an asthma diagnosis.

Exclusion Criteria:

* Children without accessible medical records

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Case studies will include subjects between the ages of 3-9 years who have had at least 2 asthma diagnoses within the last 2 years. Patients will be selected based upon their ICD9 codes for asthma. Control subjects will be age matched and without an asthma diagnosis.
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2005-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Halterman, MD, MPH, Principal Investigator — University of Rochester; Ritu Pabby, MD, Study Chair — West Penn Allegheny Health System
Locations (1):
- Department of Pediatrics, University of Rochester, Rochester, New York, United States